CLINICAL TRIAL: NCT02992379
Title: Clinical Evaluation of Stabilizing Splint Versus Pivot Splint as Jaw Exercise Together With Stabilizing Splint as Treatment for TMJ Anterior Disc Displacement Without Reduction
Brief Title: Clinical Evaluation of Stabilizing Splint Versus Pivot Splint as Jaw Exercise Together With Stabilizing Splint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hesham Mohamed mohamed elsayed safa, Resident at National Cancer Institute, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cairo ss-ps
Record Dates: First submitted 2016-11-29; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: TMJ Disc Disorder
Keywords: Anterior disc displacement; Stabilizing splint

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- stabilizing splint (Active Comparator): Active Comparator: stabilizing splint A 2-mm-thick, hard, clear sheet of resin will be adapted to the maxillary arch . Small amount of self-curing acrylic will be added to the anterior portion of the appliance as a stop for the lower incisor. The area of this stop is approximately 4 to 6 mm. The patient is instructed to protrude the mandible slightly and to open and close the mouth In this position. Self-curing acrylic will be added to the occluding surface of the appliance. All occluding areas, except the contact on the anterior stop . Excess acrylic surrounding the centric contacts is removed with a hard rubber wheel on a lathe. intervention: pivot splint
  Interventions: Device: pivot splint; Device: stabilizing splint
- pivot splint (Experimental): Experimental: pivot splint A 2-mm-thick, hard, clear sheet of resin will be adapted to the maxillary arch . Small amount of self-curing acrylic will be added to the anterior portion of the appliance as a stop for the lower incisor. The area of this stop is approximately 4 to 6 mm. The patient should be instructed to close in Centric relation . Self-curing acrylic will be added to the occluding surface of the appliance. All occluding areas, except the contact on the anterior stop . Excess acrylic surrounding the centric contacts is removed with a hard rubber wheel on a lathe. All areas, except labial to the mandibular canines, are flattened to the contact marks.
  Other Names: PS
  Interventions: Device: pivot splint; Device: stabilizing splint

INTERVENTIONS:
Device: pivot splint — A 2-mm-thick, hard, clear sheet of resin will be adapted to the maxillary arch . Small amount of selfcuring acrylic will be added to the anterior portion of the appliance as a stop for the lower incisor. The area of this stop is approximately 4 to 6 mm. The patient is instructed to protrude the mandible slightly and to open and close the mouth In this position. Self-curing acrylic will be added to the occluding surface of the appliance. All occluding areas, except the contact on the anterior stop . Excess acrylic surrounding the centric contacts is removed with a hard rubber wheel on a lathe.
  Other Names: PS
Device: stabilizing splint — A 2-mm-thick, hard, clear sheet of resin will be adapted to the maxillary arch . Small amount of self-curing acrylic will be added to the anterior portion of the appliance as a stop for the lower incisor. The area of this stop is approximately 4 to 6 mm. The patient is instructed to protrude the mandible slightly and to open and close the mouth In this position. Self-curing acrylic will be added to the occluding surface of the appliance. All occluding areas, except the contact on the anterior stop . Excess acrylic surrounding the centric contacts is removed with a hard rubber wheel on a lathe. intervention: pivot splint

SUMMARY:
To evaluate the effectiveness of the stabilizing splint versus the pivot splint as jaw exercise together with stabilizing splints for treatment of TMJ anterior disc displacement without reduction

DETAILED DESCRIPTION:
To evaluate the effectiveness of the stabilizing splint versus the pivot splint as jaw exercise together with stabilizing splints for treatment of TMJ anterior disc displacement without reduction

PICO:

Population (P): Patients with symptomatic anterior disc displacement without reduction.

Intervention (I): pivot splint.

Comparator (C): stabilizing repositioning splint (ARS).

Outcome (O):

Primary outcome:

Patients' subjective pain experience. Each patient will be asked to rate his or her current and worst pain intensity on numerical rating scale (NRS) of 0-10 with zero being no pain and ten corresponds to the worst pain that the patient ever had.

Secondary outcome:

1. Maximum mouth opening (MMO). Assessment of MMO will be performed by measuring the distance in mm between the incisal edges of the upper and lower central incisors using a ruler.
2. Lateral excursion. Assessment of lateral excursion will be performed by measuring the distance in mm between midline of upper and lower jaws
3. Protrusion. distance in mm from the incisal edge of the maxillary central incisor to the incisor edge of the mandibular incisor will measured in the maximum protruded position.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient from 15 to 50 years old
* Report of pain in preauricular region worsened by functional activities, such as chewing and talking
* Presence of disc displacement with reduction and joint clicking
* Positive diagnosis of unilateral or bilateral anterior disc displacement with reduction by means of magnetic resonance imaging (MRI)

Exclusion Criteria:

* Individuals with systemic diseases that can affect TMJ
* History of TMJ surgery
* Individuals with osteoarthritis
* Individuals under TMD management
* Individuals wearing full or partial dentures
* Reducing dislocations of the articular disc
* Consequences of condyle fractures and/or fracture of another maxillofacial zone
* In therapy for the same pathologies
* Articular pathologies of systemic nature (e.g., rheumatoid arthritis, arthrosis, psoriasis arthritis)
* Individuals with a recent history of trauma in the face and/or neck area

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Patients' subjective pain experience (numerical rating scale) | 6 months
  Each patient will be asked to rate his or her current and worst pain intensity on numerical rating scale (NRS) of 0-10 with zero being no pain and ten corresponds to the worst pain that the patient ever had.

SECONDARY OUTCOMES:
Maximum mouth opening (Unit: mm) | 6 months
  measuring the distance between the incisal edges of the upper and lower central incisors using a ruler. Unit: mm
Lateral excursion (Unit: mm) | 6 months
  measuring the distance between midline of upper and lower jaws. Unit: mm
Protrusion (distance in mm) | 6 months
  The distance in mm from the incisal edge of the maxillary central incisor to the incisor edge of the mandibular incisor will measured in the maximum protruded position.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Galal, Ass.prof, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ebrahim S, Montoya L, Busse JW, Carrasco-Labra A, Guyatt GH; Medically Unexplained Syndromes Research Group. The effectiveness of splint therapy in patients with temporomandibular disorders: a systematic review and meta-analysis. J Am Dent Assoc. 2012 Aug;143(8):847-57. doi: 10.14219/jada.archive.2012.0289. PMID 22855899